CLINICAL TRIAL: NCT03827941
Title: Auricular Transcutaneous Electrical Nerve Stimulation Treatment of Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P000894
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 Hz group (Active Comparator): 1 Hz Auricular transcutaneous electrical nerve stimulation High-functioning individuals with autism randomized to this group will receive 1 Hz tVNS stimulation for 30 minutes/day up to 5 times/week for 3 weeks.
  Interventions: Other: 1 Hz Auricular transcutaneous electrical nerve stimulation
- 20 Hz group (Active Comparator): 20 Hz Auricular transcutaneous electrical nerve stimulation High-functioning individuals with autism randomized to this group will receive 20 Hz tVNS stimulation for 30 minutes/day up to 5 times/week for 3 weeks.
  Interventions: Other: 20 Hz Auricular transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: 1 Hz Auricular transcutaneous electrical nerve stimulation — High-functioning individuals with autism randomized to this group will receive 1 Hz tVNS stimulation for 30 minutes/day up to 5 times/week for 3 weeks.
  Arms: 1 Hz group
Other: 20 Hz Auricular transcutaneous electrical nerve stimulation — High-functioning individuals with autism randomized to this group will receive 1 Hz tVNS stimulation for 30 minutes/day up to 5 times/week for 3 weeks.
  Arms: 20 Hz group

SUMMARY:
In this study, investigators will examine the treatment effects of transcutaneous electrical nerve stimulation with different stimulation frequencies on individuals with autism.

DETAILED DESCRIPTION:
In this study, investigators will examine the treatment effect of transcutaneous electrical nerve stimulation at auricular area with vagus nerve distribution on high-functioning individuals with autism. Specifically, investigators will choose two ear acupoints: heart and shenmen. Participants will be randomized to either 1 Hz or 20 Hz tVNS group (up to 5 times per week) for three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Autism diagnosed based on DSM-V classification criteria
2. 18-60 year old high functioning adult autism patients (e.g. Asperger's, IQ equal or greater than 80)
3. Subjects who do not show aggressive behaviors based on neuro/psychiatric evaluations as determined by a licensed study physician.

Exclusion Criteria:

1. A history of chronic serious infection, any current infection, any type of cancer or autoimmune disease or other severe diseases;
2. Subjects taking any medications that confound the study results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-01-28 (Estimated); Study Completion 2024-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in Autism Treatment Evaluation Checklist (ATEC) | Baseline and after 3-week treatment
  ATEC will be reported by investigator in a total and for each of the 4 subscales as follows: (1) speech/language/communication subscale; (2) social subscale; (3) sensory and cognitive awareness subscale; and (4) health / physical / behavior problem subscale. The total score ranges from 0 to 179; a higher score indicated worsening while a lower score indicated improvement.

SECONDARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) | Baseline and after 3-week treatment
  The factors of the ABC have been labeled as follows: (I) Irritability, Agitation, Crying; (II) Lethargy, Social Withdrawal; (III) Stereotypic Behavior; (IV) Hyperactivity, Noncompliance; and (V) Inappropriate Speech.
Change in Clinical Global Impression-Improvement (CGI-I) | Baseline and after 3-week treatment
  Overall improvement in autism will be assessed using the Clinical Global Impression-Improvement (CGI-I) scale, a 7-point scale from 1 = very much improved to 7 = very much worse.
Change in PROMIS Sleep Disturbance Short Form | Baseline and after 3-week treatment
  This questionnaire is used to assess the pure domain of sleep disturbance in adults.
Change in Penn State Worry Questionnaire | Baseline and after 3-week treatment
  This is the standard assessment of worry and consists of 16 questions rated from 1 to 5 from "Not typical of me" to "Very typical of me".
Change in Sleep Quality Assessment (PSQI) | Baseline and after 3-week treatment
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last week.
PROMIS-29 | Baseline and after 3-week treatment
  The PROMIS-29 assesses pain intensity, physical function, depression, anxiety, fatigue, sleep disturbance, interference, and social role and activity in the past 7 days
EEG (optional) | Baseline and after 3-week treatment
  Resting state EEG (filter 1-50 Hz) will be collected
Salivary oxytocin quantification (optional) | Baseline and after 3-week treatment
  A total of 4-mL of unstimulated saliva will be collected
Quantification of species-level L. reuteri abundance in human stool samples (optional) | Baseline and after 3-week treatment
  Stool samples will be collected at home following our provided instructions.
Autonomic measurements via wristband photoplethysmograph (PPG) sensor (optional) | Baseline and after 3-week treatment
  6 minutes PPG data will be collected
ECG (optional) | Baseline and after 3-week treatment
  6 minutes raw ECG data will be collected for Heart rate variability (HRV) analysis
Pulse oximetry measurements (optional) | Baseline and after 3-week treatment
  SpCO will be measured at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, Principal Investigator — MGH

IPD SHARING:
Plan to Share IPD: No